CLINICAL TRIAL: NCT03514329
Title: Vapor Ablation for Localized Cancer Lesions of the Lung - A Clinical Feasibility Definitive Treatment Study
Brief Title: Vapor Ablation for Localized Cancer Lesions
Acronym: VAPORIZED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uptake Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-2315
Record Dates: First submitted 2017-09-25; First posted 2018-05-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer; Metastatic Lung Cancer; Lung Cancer
Keywords: Non Small Cell Lung Cancer; Metastatic Lung Cancer; Lung Cancer; Vapor Ablation; BTVA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vapor Ablation (Experimental): Patients treated with Bronchoscopic Thermal Vapor Ablation for lung cancer
  Interventions: Device: Bronchoscopic Thermal Vapor Ablation

INTERVENTIONS:
Device: Bronchoscopic Thermal Vapor Ablation — Vapor (steam) is infused into the targeted region for 8 seconds at a precisely controlled flow rate and power.
  Other Names: BTVA-C

SUMMARY:
This study is a prospective, single-arm, multi-center, pilot trial of Bronchoscopic Thermal Vapor Ablation for Lung Cancer (BTVA-C) in patients with primary lung cancer or metastatic cancer in the lung. Patients who have consented to participate in this study (enrolled) will be subject to eligibility screening and baseline assessments, prior to undergoing the BTVA-C procedure. Only patients that meet all of the inclusion criteria and none of the exclusion criteria will receive vapor ablation treatment.

Patients will be followed for up to 12 months.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multi-center, pilot trial of Bronchoscopic Thermal Vapor Ablation for Lung Cancer (BTVA-C) in patients with primary lung cancer or metastatic cancer in the lung.

Subjects identified for this study will be those that have microscopic proof of malignancy. Patients who have consented to participate in this study (enrolled) will undergo screening assessments to evaluate the inclusion criteria associated with their lung cancer and general health. Only patients that meet all of the inclusion criteria and none of the exclusion criteria will be scheduled for treatment with the BTAV-C System.

A total of 10 subjects will be treated at up to 3 investigational sites within the EU.

Prior to the vapor ablation procedure, the patient's CT scan is analyzed to evaluate the location and size of the target lesion. The segments and airways associated with the lesion are identified and images are created to aid in the navigation to appropriate treatment locations during the upcoming procedure.

At the time of the vapor ablation procedure, the Uptake catheter is placed in a selected airway with a thin bronchoscope. A balloon at the distal end of the catheter is then inflated to occlude the bronchus prior to vapor infusion. Sterile water is heated to approximately 100° - 140°C by a reusable generator and vapor (steam) is infused into the targeted region for 8 seconds at a precisely controlled flow rate and power. If necessary, the catheter is moved to the next airway and the procedure is repeated until all desired airways have been treated (maximum 3 treatments). The treatment creates a uniform field of necrosis in the parenchyma around the lesion.

Patients will be evaluated for clinical symptoms in the 30-day period following ablation. Local control of the tumor will be evaluated based on Response Evaluation Criteria in Solid Tumors (RECIST) from low dose CT scans at 1, 3, 6 and 12 months following ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old
2. Patient has been recommended for ablation or recommended for an alternative to surgery
3. Non-small cell lung cancer tumor(s) ≤ 2cm (T1aN0, T1bN0) OR Metastatic lung tumor(s) ≤ 2cm
4. Microscopic proof of malignancy obtained
5. Location of tumor:

   1. In periphery of lung (outermost 1/3)
   2. Maximum of three vapor ablation applications would target entire margin according to the vapor ablation plan
6. Signed patient informed consent

Exclusion Criteria:

1. Centralized tumor (abutting main stem bronchus, main pulmonary artery branches, esophagus, or trachea)
2. Carcinoid lung tumors
3. Tumor is associated with atelectasis or obstructive pneumonitis or pleural effusion
4. Pulmonary function tests (PFTs): post-bronchodilator forced expired volume in one second (FEV1) <20% predicted, diffusing capacity of the lung for carbon monoxide (DLCO)<20% predicted
5. Requirement for supplemental oxygen (includes at rest or during exercise)
6. Hospitalization for cardiac disease within the preceding 6 months
7. Liver enzymes (ALP, ALT, AST) or total bilirubin > 1.5 upper limit of normal (ULN)
8. Serum creatinine > 2 mg/dl
9. Recent infection (within 30 days)
10. Currently receiving immunosuppressive medication or prednisone > 10 mg/day (or equivalent)
11. Pre-existing implants within the airways that impede navigation to the target lesion
12. Pregnant or breastfeeding women and those of childbearing potential who are not practicing a reliable form of contraception.
13. Disorder of coagulation, history of severe hemoptysis, or receiving anticoagulant medication. Antiplatelet medication is permitted provided that the medication can be held a minimum of 7 days prior to the procedure and 10 days post-procedure.
14. Any condition that in the opinion of the investigator or reviewer may interfere with the safety of the patient or evaluation of the study objectives
15. Any tumor characteristic that in the opinion of the investigator or reviewers may interfere with the safety of the patient or evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
BTVA-C related AEs/SAEs | up to 6 months post-ablation
  The number of reported adverse events (AEs), serious adverse events (SAEs) related to the BTVA-C procedure.
Successful BTVA-C Treatment Delivery | Day 0
  Treatment meets 100% of the required procedural steps/requirements per the Instructions for Use (IFU) and treatment is delivered to the target tumor per the individual patient navigation plan
Local Control Evaluation per RECIST | Month 1, 3, 6, and 12
  Evaluation in the change in response to vapor ablation based on the RECIST 1.1 protocol

CONTACTS AND LOCATIONS:
Locations (2):
- Otto-Wagner Hospital, Vienna, Austria
- Azienda Ospedaliero - Universitaria, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Uptake Medical website — http://www.uptakemedical.com/